CLINICAL TRIAL: NCT05819632
Title: Clinical Comparison of Topical Application of Curcumin Gel Versus Gelatin Sponge in Pain Management and Wound Healing After Free Gingival Graft Harvesting: a Randomized Controlled Clinical Trial
Brief Title: Clinical Comparison of Application of Curcumin Gel in Pain Management After Free Gingival Graft Harvesting
Acronym: curcumin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tansim Khaled Tawfik Abdelrahman, masters degree candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CairoU28122022
Record Dates: First submitted 2023-03-03; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Palate; Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- curcumin gel (Experimental): the denuded palatal area will be superficially covered with a continuous thin layer of curcumin gel 2% one time immediately after the surgery (curcumin gel will be prepared in 2% concentration on a carbapol base)according to (Bhatia et al., 2014)
  Interventions: Other: curcumin gel 2%
- gelatine sponge (Active Comparator): absorbable gelatin sponge will be cut to the palatal wound size and applied. Following manual compression of the wound area, both agents will be secured in place using compressive palatal sling sutures.
  commercial name (CUTANPLAST)
  Interventions: Other: curcumin gel 2%

INTERVENTIONS:
Other: curcumin gel 2% — curcumin gel 2%

SUMMARY:
The aim of this study is to compare the effect of using 2% curcumin gel versus gelatin sponge when applied to palatal donor site in pain management and wound healing after free gingival graft harvesting.

ELIGIBILITY:
Inclusion Criteria:

1. Systematically healthy patient (American Society of Anesthesiology class I and II).
2. Male or female
3. Patients with mucogingival defects scheduled for free gingival graft.
4. Patients with good oral hygiene.

Exclusion Criteria:

1. Patients with any uncontrolled local or systemic disease where periodontal plastic surgery might be contraindicated.
2. History of recent periodontal surgery at the donor site.
3. Smokers.
4. Pregnancy and lactation.
5. Patients allergic to the used agents,
6. Severe gagging reflex.
7. Inability or unwillingness to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
post-operative pain | one week post operative
  post -operative pain measured by visual analouge scale from 0 (no pain) to 10 (highest pain value)

SECONDARY OUTCOMES:
Soft tissue healing of the palatal wound | up to three weeks post-operative
  Soft tissue healing of the palatal wound measured by Modified Landry's wound healing score from 1 indicates poorest healing to 5 indicates excellent healing
Re-epithelization of the palatal wound | up to three weeks post-operative
  Re-epithelization of the palatal wound using H2O2 test

CONTACTS AND LOCATIONS:
Overall Officials: tansim k abdelrahman, BDS, Principal Investigator — master student; mohamed Atef, PHD, Study Director — Lecture of oral medicine and periodontology, faculty of dentistry ,Cairo university; manal m hosny, phd, Study Chair — Professor of oral medicine and periodontology factuality of Dentistry,Cairo university
Locations (1):
- Faculty of Dentistry, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No